CLINICAL TRIAL: NCT06189092
Title: Trattamento Delle Malformazioni Venose a Basso Flusso Con l'Elettroscleroterapia. Studio Osservazionale Prospettico
Brief Title: Treatment of Low-flow Venous Malformations With Electrosclerotherapy. Prospective Observational Study
Acronym: BESVAM
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC: 639/2023/Oss/IOR
Record Dates: First submitted 2023-11-30; First posted 2024-01-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Vascular Malformations
Keywords: Electrosclerotherapy
MeSH Terms: conditions — Vascular Malformations | interventions — Bleomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Performed electrosclerotherapy: All patients who performed electrosclerotherapy in the treatment of vascular malformations
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin — Using electroporation to infuse bleomycin in the lesion

SUMMARY:
Venous malformations (MVs) are congenital abnormalities of the central or periphery caused by developmental errors at different stages of embryogenesis. Histologically they are characterized by large, venous-like vascular spaces. Scleroembolization constitutes the most widespread method in the treatment of venous malformations allowing good results with low invasiveness. Currently, Bleomycin (and its derivatives) is among the most widely used sclerosing agents for slow-flowing vascular malformations (venous and lymphatic malformations) because of the low rate of local serious adverse events such as swelling, necrosis, and nerve injury compared with others.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of low-flow venous malformations eligible for electrosclerotherapy
* Non-indication for embolizing treatment
* Previous treatments are not an exclusion factor, provided that at least 30 days have elapsed.

Exclusion Criteria:

* Previous treatment for < 30 days
* Pregnancy and lactation status
* Patients of childbearing age without contraceptive use
* Presence of metal synthetic media
* COPD with FiO2 < 30 mmHg
* Impaired renal function with eGFR<30 ml/min/1.73mq
* Patients with Bleomycin intolerance or previous episodes of toxicity Bleomycin-related
* Patients who have already received a cumulative dose of Bleomycin ≥100 mg
* Patients who have undergone prior thoracic radiotherapy
* Patients with a history of seizures and epilepsy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by low-flow vascular malformations
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
Volume reduction in cm | 1 year
  Reduction of the lesion of at least 30% evaluated with MRI, measuring the diameter of the lesion in cm.

SECONDARY OUTCOMES:
Reduction of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.
Improvement in quality of life ( EuroQol-5D questionnaire) | 1 year
  Clinical assessment regarding quality of life by EuroQol-5D questionnaire. EQ-5D score can range from -0.594 to 1.0.
  The minimum value represents the worst possible health condition. The maximum value of 1.0 represents the best possible health condition. A value of 1.0 indicates that the patient has no problem in any of the five dimensions assessed by the questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy